CLINICAL TRIAL: NCT05043077
Title: Efficacy and Safety of Mydriatic Microdrops for Retinopathy Of Prematurity Screening: a Non-inferiority Crossover Randomized Controlled Trial (MyMiROPS Trial)
Brief Title: Efficacy and Safety of Mydriatic Microdrops for Retinopathy Of Prematurity Screening
Acronym: MyMiROPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Asimina Mataftsi, Associate Professor in Ophthalmology, Paediatric Ophthalmology and Strabismus, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Screening
Other Study IDs: 23265/14-07-2021
Record Dates: First submitted 2021-09-02; First posted 2021-09-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Retinopathy of Prematurity
Keywords: microdrops; mydriasis; dilating drops; phenylephrine; tropicamide; retinopathy of prematurity; ROP; screening
MeSH Terms: conditions — Retinopathy of Prematurity; Mydriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Mydriasis with microdrops
  Interventions: Drug: Microdrop administration of phenylephrine 1.67% and tropicamide 0.33%
- Control Group (Active Comparator): Mydriasis with standard drops
  Interventions: Drug: Standard drop administration of phenylephrine 1.67% and tropicamide 0.33%

INTERVENTIONS:
Drug: Microdrop administration of phenylephrine 1.67% and tropicamide 0.33% — 1 drop (6.5 μL) for 3 doses with 5-minute intervals
  Arms: Study Group
Drug: Standard drop administration of phenylephrine 1.67% and tropicamide 0.33% — 1 drop (28-34 μL) for 3 doses with 5-minute intervals
  Arms: Control Group

SUMMARY:
The purpose is to test the hypothesis that microdrop instillation of combined phenylephrine 1.67% and tropicamide 0.33% eyedrops causes at least equal mydriasis compared with standard drop instillation of the same mydriatic regimen, which constitutes routine care for pupil dilation during retinopathy of prematurity (ROP) screening in our neonatal intensive care unit. Comparison, also, will be made to the subsequent adverse events and the drug concentration in peripheral blood samples.

DETAILED DESCRIPTION:
A non-inferiority, crossover, randomized controlled trial will be conducted for this purpose. Participants will be randomly assigned to receive either a) microdrops on their first and standard drops on their second screening examination a week later (M/S group), or b) standard drops first and microdrops a week later (S/M group). Microdrops (6.5 μL) will be instilled using a calibrated micropipette, while standard drops (28-34 μL) will be instilled directly through the commercially available plastic multi-dose mydriatic dropper bottle.

ELIGIBILITY:
Inclusion Criteria:

Preterm infants undergoing screening for ROP, i.e.

* infants with GA < 32 weeks and/or BW < 1501 grams
* infants of greater GA and BW with comorbidities, e.g. sepsis, prolonged need for oxygen supplementation etc., as recommended by the attending neonatologist

Exclusion Criteria:

* Unstable clinical condition
* Severe cardiovascular disease
* Congenital anomalies
* Clinical syndromes
* Inotropes' intake during the week prior to enrollment
* Traumatic apoptosis of the corneal epithelium
* Corneal ulcer
* Anatomical variations of the anterior segment
* Infants that are outpatients at the commencement of ROP screening

Ages: 30 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Mydriatic efficacy: millimeters of horizontal pupil diameter. | 45 minutes after the first drop instillation.

SECONDARY OUTCOMES:
Mydriasis sustainability: millimeters of horizontal pupil diameter. | 90 minutes after the first drop instillation.
Mydriasis sustainability: millimeters of horizontal pupil diameter. | 120 minutes after the first drop instillation.
Pharmacokinetic profile of phenylephrine: area under the whole blood concentration versus time curve (AUC). | Blood sampling at 15, 20, 25, 30, 40, 50, 60, 120, and 180 minutes after the first drop instillation.
  Each participant will be sampled once (random allocation to one time-point). Blood sampling will be combined with peripheral blood collection for routine examinations.
Pharmacokinetic profile of phenylephrine: maximum (peak) whole blood concentration (Cmax). | Blood sampling at 15, 20, 25, 30, 40, 50, 60, 120, and 180 minutes after the first drop instillation.
  Each participant will be sampled once (random allocation to one time-point). Blood sampling will be combined with peripheral blood collection for routine examinations.
Pharmacokinetic profile of phenylephrine: time to reach maximum (peak) whole blood concentration (Tmax). | Blood sampling at 15, 20, 25, 30, 40, 50, 60, 120, and 180 minutes after the first drop instillation.
  Each participant will be sampled once (random allocation to one time-point). Blood sampling will be combined with peripheral blood collection for routine examinations.
Pharmacokinetic profile of phenylephrine: elimination half-life (T1/2). | Blood sampling at 15, 20, 25, 30, 40, 50, 60, 120, and 180 minutes after the first drop instillation.
  Each participant will be sampled once (random allocation to one time-point). Blood sampling will be combined with peripheral blood collection for routine examinations.
Heart rate values (beats per minute). | 45, 90 and 120 minutes after the first drop instillation.
Oxygen saturation (SpO2) values (%). | 45, 90 and 120 minutes after the first drop instillation.
Systolic, diastolic, and mean blood pressure values (mmHg). | 45, 90 and 120 minutes after the first drop instillation. Hourly blood pressure measurements for the first 24 hours after mydriasis.
Number of participants with systemic adverse events. | During the 48 hours after mydriasis.
  Apnea, increased gastric residuals, inhibited duodenal motor activity, delayed gastric emptying, feeding intolerance, abdominal distension, vomiting, paralytic ileus, acute gastric dilatation, necrotizing enterocolitis (NEC).
Number of participants with local adverse events. | 45 minutes after the first drop instillation.
  Periorbital pallor, eyelid swelling, flushing.
Adequacy of judging the presence or absence of treatment-requiring ROP. | At the end of the eye examination (fundoscopy).

CONTACTS AND LOCATIONS:
Locations (1):
- Papageorgiou General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes
Deidentified Individual Participant Data (IPD) that underline published results, along with related data dictionaries, will be available from 3 months to 36 months following article publication, only to researchers who will provide a methodologically sound proposal, for types of analyses to achieve aims in the approved proposal or for individual participant data meta-analysis, and only after acceptance of the proposed protocol by our Institution's IRB. Proposals should be directed to the corresponding author (AM, amatafts@auth.gr) and data requestors will need to sign a data access agreement. The study protocol and statistical analysis plan will also be available, if needed.

REFERENCES:
- [Background] Lynch MG, Brown RH, Goode SM, Schoenwald RD, Chien DS. Reduction of phenylephrine drop size in infants achieves equal dilation with decreased systemic absorption. Arch Ophthalmol. 1987 Oct;105(10):1364-5. doi: 10.1001/archopht.1987.01060100066027. PMID 3662909
- [Background] Elibol O, Alcelik T, Yuksel N, Caglar Y. The influence of drop size of cyclopentolate, phenylephrine and tropicamide on pupil dilatation and systemic side effects in infants. Acta Ophthalmol Scand. 1997 Apr;75(2):178-80. doi: 10.1111/j.1600-0420.1997.tb00119.x. PMID 9197568
- [Background] Seliniotaki AK, Prousali E, Lithoxopoulou M, Kokkali S, Ziakas N, Soubasi V, Mataftsi A. Alternative mydriasis techniques for retinopathy of prematurity screening. Int Ophthalmol. 2020 Dec;40(12):3613-3619. doi: 10.1007/s10792-020-01542-x. Epub 2020 Aug 9. PMID 32772218
- [Result] Seliniotaki AK, Lithoxopoulou M, Virgiliou C, Gika H, Dokoumetzidis A, Bougioukas KI, Raikos N, Diamanti E, Ziakas N, Haidich AB, Mataftsi A. Efficacy and Safety of Mydriatic Microdrops for Retinopathy of Prematurity Screening: The MyMiROPS Randomized Clinical Trial. JAMA Ophthalmol. 2025 Feb 1;143(2):110-116. doi: 10.1001/jamaophthalmol.2024.5462. PMID 39724200
- [Derived] Seliniotaki AK, Haidich AB, Lithoxopoulou M, Gika H, Boutou E, Virgiliou C, Nikolaidou M, Dokoumetzidis A, Raikos N, Diamanti E, Ziakas N, Mataftsi A. Efficacy and safety of Mydriatic Microdrops for Retinopathy Of Prematurity Screening (MyMiROPS): study protocol for a non-inferiority crossover randomized controlled trial. Trials. 2022 Apr 15;23(1):322. doi: 10.1186/s13063-022-06243-7. PMID 35428316